CLINICAL TRIAL: NCT03060395
Title: Effects of A2 Milk on Gastrointestinal Function of Volunteers Affected by Non-lactose Milk Intolerance
Brief Title: Effects of A2 Milk on Gastrointestinal Function in Non-lactose Milk Intolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Sandrine Claus, Associate Professor in Integrative Metabolism, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: A2study
Record Dates: First submitted 2017-01-17; First posted 2017-02-23 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Milk Intolerance
MeSH Terms: conditions — Lactose Intolerance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A1/A2 milk (Sham Comparator): Commercial conventional A1/A2 semi-skimmed fresh pasteurised cow milk. Progressive intake of intervention milk as follows:
  * Days 1 and 2: 100 mL twice a day
  * Days 3 and 4: 150 mL twice a day
  * Days 5 and 6: 200 mL twice a day
  * Days 7 to 14: 250 mL twice a day
  Interventions: Dietary Supplement: A1/A2 milk 100; Dietary Supplement: A1/A2 milk 150; Dietary Supplement: A1/A2 milk 200; Dietary Supplement: A1/A2 milk 250
- A2 milk (Active Comparator): Commercial A2 semi-skimmed fresh pasteurised cow milk.
  Progressive intake of intervention milk as follows:
  * Days 1 and 2: 100 mL twice a day
  * Days 3 and 4: 150 mL twice a day
  * Days 5 and 6: 200 mL twice a day
  * Days 7 to 14: 250 mL twice a day
  Interventions: Dietary Supplement: A2 milk 100; Dietary Supplement: A2 milk 150; Dietary Supplement: A2 milk 200; Dietary Supplement: A2 milk 250

INTERVENTIONS:
Dietary Supplement: A2 milk 100 — Days 1 and 2: 100 mL A2 milk twice a day
  Arms: A2 milk
Dietary Supplement: A2 milk 150 — Days 3 and 4: 150 mL A2 milk twice a day
  Arms: A2 milk
Dietary Supplement: A2 milk 200 — Days 5 and 6: 200 mL A2 milk twice a day
  Arms: A2 milk
Dietary Supplement: A2 milk 250 — Days 7 to 14: 250 mL A2 milk twice a day
  Arms: A2 milk
Dietary Supplement: A1/A2 milk 100 — Days 1 and 2: 100 mL A1/A2 milk twice a day
  Arms: A1/A2 milk
Dietary Supplement: A1/A2 milk 150 — Days 3 and 4: 150 mL A1/A2 milk twice a day
  Arms: A1/A2 milk
Dietary Supplement: A1/A2 milk 200 — Days 5 and 6: 200 mL A1/A2 milk twice a day
  Arms: A1/A2 milk
Dietary Supplement: A1/A2 milk 250 — Days 7 to14: 250 mL A1/A2 milk twice a day
  Arms: A1/A2 milk

SUMMARY:
There is increasing evidence that a number of people experience moderate milk intolerance characterised by increased gas production, bloating and abdominal cramp, which can neither be attributed to lactose intolerance, nor to milk protein allergy. Milk digestion can lead to the formation of bioactive peptides, one of which derived from a mutated gene variant (A1) coding for milk beta-casein has been associated with increased gastrointestinal inflammation and poor gastrointestinal function. In this study, we hypothesise that consumption of non-mutated A2 milk will improve gastrointestinal symptoms in non-lactose milk intolerant individuals.

DETAILED DESCRIPTION:
Non-lactose milk intolerance is a condition that has not been defined clinically yet but the current literature reports existence of subjects who are moderately milk intolerant and whose intolerance can neither be attributed to a defect in lactose intolerance, nor to milk protein allergy. Yet, they experience at least one or two of the following symptoms following milk consumption: gases, bloating, abdominal cramp. It is known that the A1gene variant coding for beta-casein leads to the production of a bioactive peptide with opioid activity named betacasomorphin 7 (BCM7). This peptide has been associated with several metabolic health disorders including diabetes, elevated cardiovascular risk and stimulation of pro-inflammatory signals. Recently, it was reported that non-lactose milk intolerant subjects did not experience such symptoms when consuming milk containing the non-mutated A2 gene variant coding for beta-casein. In this study, we hypothesise that consumption of A2 milk will improve gastrointestinal symptoms in non-lactose milk intolerant individuals. The primary outcome of this study will be the reduction of gastrointestinal inflammation following a course of A2 milk consumption.

ELIGIBILITY:
Inclusion Criteria:

* BMI: 20-35kg/m2
* Glucose<7mmol/l (not diagnosed with diabetes)
* Total cholesterol<7mmol/l
* Triacylglycerol<4mmol/l
* Normal liver and kidney function
* Regular milk drinker with self-reported intolerance to commercial milk.
* Suffered from mild to moderate digestive discomfort after milk consumption.
* Have normal blood pressure 120/80 mmHg (BP <160/90 mmHg can be accepted) during quiet respiration.
* Agree not to take any medication, supplements and other dairy products including acidophilus milk
* Be willing to comply with all the requirements and procedures of the study.
* Agree to sign the informed consent form;
* Agree not to enrol in another interventional clinical research study while participating in this study.
* Fully understand the nature, objective, benefit and the potential risks and side effects of the study.

Exclusion Criteria:

* Females who are pregnant or planning to be a pregnant and lactating.
* Have known dairy allergy.
* Have stopped drinking milk for the last 6 month.
* Have history of lactose intolerance
* Have history of faecal impaction.
* Received antibiotics in the previous six months
* Smoker
* Anemia
* Trying to lose weight by following a diet or exercise regimen designed for weight loss, or taking any drug influencing appetite and any drug for weight loss for the last three months.
* Have participated in similar dairy or probiotics-containing product's clinical trials within 3 months before the screening.
* Currently taking medicines for cardiovascular or metabolic disease.
* History of alcohol or drug misuse.
* Have history of or be diagnosed of any of the following diseases that may affect the study results: gastrointestinal disorders, hepatopathy, nephropathy, endocrine disease, blood disorders, respiratory, cardiovascular diseases and known on-going allergy such as asthma.
* Currently suffering from any gastrointestinal disorders or gastrointestinal disease, including irritable bowel syndrome, colitis, ulcerative colitis, celiac disease, irritable bowel syndrome (IBS);
* Had hospitalizations within 3 months before screening; Currently drug frequency user of that may affect the gastrointestinal function or immune system. As judged by investigator.
* Who take medication at least the last 6-month.
* Who do excessive exercise not as part of a weight-loss regime, e.g. athletes.

Ages: 18 Years to 56 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Change in gastrointestinal inflammation indicated by fecal calprotectin | baseline, 14 days, 28 days, 42 days and 56 days
  Measurement of fecal calprotectin (ug/g feces)

SECONDARY OUTCOMES:
Change in NMR-based urinary metabolic profiles | baseline, 14 days, 28 days, 42 days and 56 days
  Measured using High Resolution 700MHz proton NMR spectroscopy (Bruker) (no unit)
Change in NMR-based plasma metabolic profiles | baseline, 14 days, 28 days, 42 days and 56 days
  Measured using High Resolution 700MHz proton NMR spectroscopy (Bruker) (no unit)
Change in NMR-based fecal metabolic profiles | baseline, 14 days, 28 days, 42 days and 56 days
  Measured using High Resolution 700MHz proton NMR spectroscopy (Bruker) (no unit)
Change in gut microbiota ecosystem assessed by sequencing the 16S rDNA extracted from feces | baseline, 14 days, 28 days, 42 days and 56 days
  Measures relative abundance of bacterial taxa
Change in systemic inflammation indicated by circulating levels of high sensitivity C-reactive protein | baseline, 14 days, 28 days, 42 days and 56 days
  hs-CRP in mg/L
Change in gastrointestinal function assessed using visual analogue scale for GI symptoms | 14 days
  Measures gases, bloating, abdominal cramps, diarrhoea, headache, constipation, nausea and rash
Height (in m) used to detect change in BMI (kg/m^2) | baseline
Weight (in kg) used to detect change in BMI (kg/m^2) | baseline, 14 days, 28 days, 42 days and 56 days
Change in systolic blood pressure in mmHg | baseline, 14 days, 28 days, 42 days and 56 days
Change in diastolic blood pressure in mmHg | baseline, 14 days, 28 days, 42 days and 56 days
Diagnostic of lactose intolerance by breath hydrogen concentration following ingestion of 25g lactose in 250 mL water | screening visit, 14 days, 42 days and 56 days
Diagnostic of lactose intolerance by breath methane concentration following ingestion of 25g lactose in 250 mL water | screening visit, 14 days, 42 days and 56 days
Self-reported change in gut transit time | 14 days, 42 days and 56 days
Monitoring of changes in psychological behaviour assessed by TMT | baseline, 14 days, 28 days, 42 days and 56 days
Monitoring of changes in psychological behaviour assessed by Letter Memory Test | baseline, 14 days, 28 days, 42 days and 56 days
Monitoring of changes in psychological behaviour assessed by Flanger Test | baseline, 14 days, 28 days, 42 days and 56 days
Monitoring of changes in mood measured by PANAS questionnaire | baseline, 14 days, 28 days, 42 days and 56 days
Change in stool consistency using the Bristol stool chart | baseline, 14 days, 28 days, 42 days and 56 days

CONTACTS AND LOCATIONS:
Overall Officials: Sandrine P Claus, PhD, Principal Investigator — University of Reading
Locations (1):
- Department of Food and Nutritional Sciences, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We do not plan to share IPD with other researchers outside the University of Reading. Anonymous data may be made available upon publication of the study outcome in appropriate repositories (e.g. metabolomic profiles).

REFERENCES:
- [Background] Ul Haq MR, Kapila R, Sharma R, Saliganti V, Kapila S. Comparative evaluation of cow beta-casein variants (A1/A2) consumption on Th2-mediated inflammatory response in mouse gut. Eur J Nutr. 2014 Jun;53(4):1039-49. doi: 10.1007/s00394-013-0606-7. Epub 2013 Oct 29. PMID 24166511
- [Background] Ho S, Woodford K, Kukuljan S, Pal S. Comparative effects of A1 versus A2 beta-casein on gastrointestinal measures: a blinded randomised cross-over pilot study. Eur J Clin Nutr. 2014 Sep;68(9):994-1000. doi: 10.1038/ejcn.2014.127. Epub 2014 Jul 2. PMID 24986816
- [Background] Jianqin S, Leiming X, Lu X, Yelland GW, Ni J, Clarke AJ. Effects of milk containing only A2 beta casein versus milk containing both A1 and A2 beta casein proteins on gastrointestinal physiology, symptoms of discomfort, and cognitive behavior of people with self-reported intolerance to traditional cows' milk. Nutr J. 2016 Apr 2;15:35. doi: 10.1186/s12937-016-0147-z. PMID 27039383
- [Background] Johnson AO, Semenya JG, Buchowski MS, Enwonwu CO, Scrimshaw NS. Correlation of lactose maldigestion, lactose intolerance, and milk intolerance. Am J Clin Nutr. 1993 Mar;57(3):399-401. doi: 10.1093/ajcn/57.3.399. PMID 8438774